CLINICAL TRIAL: NCT07122206
Title: Monitoring the Response of Combination Ursodiol and Seladelpar Treatment in Primary Biliary Cholangitis Using Invasive Markers
Brief Title: Monitoring the Response of Combination Ursodiol and Seladelpar Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 031.HEP.2024.D
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Primary Biliary Cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Blood Draws — Research-related blood draws will be used to ascertain FGF19 levels.

SUMMARY:
This study aims to provide comprehensive insights into the therapeutic effects of combination treatment with ursodiol and seladelpar in PBC patients by assessing biochemical responses using biomarkers such as ALP and total bilirubin.

DETAILED DESCRIPTION:
By focusing on invasive markers like aspartate aminotransferase to platelet ratio index (APRI), enhanced liver fibrosis (ELF), 7-hydroxy-4-cholesten-3-one (C4), and fibroblast growth factor 19 (FGF19), the study will help understand the multifaceted impact of the treatment on liver fibrosis, extracellular matrix turnover, inflammation, and bile acid metabolism. This approach will ultimately guide better clinical management of PBC, allowing for tailored treatment strategies and improved patient outcomes.

The objective of this study is to evaluate the effectiveness of combined ursodiol and seladelpar treatment in PBC patients by monitoring changes in APRI, ELF score, and FGF19 levels, and validate results using traditional methods over 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis PBC as per established diagnostic criteria.
* Adults aged 18 years and older.
* Patients undergoing treatment with ursodiol (ursodeoxycholic acid) for PBC or who demonstrate intolerance to ursodiol due to side effects and persistent ALP > normal.
* Patients undergoing treatment with seladelpar for PBC.
* Patients must be willing and able to provide written informed consent for participation in the study.

Exclusion Criteria:

* Patients that do not meet inclusion criteria.
* Patients with other chronic liver diseases, such as hepatitis B, hepatitis C, non-alcoholic steatohepatitis (NASH), alcoholic liver disease, or other autoimmune liver diseases.
* Patients who have undergone a liver transplant.
* Presence of cirrhosis or hepatic decompensation at the time of study enrollment.
* Patients with significant comorbid conditions that may interfere with the study outcomes, such as severe cardiovascular, renal, or pulmonary diseases.
* Pregnant or breastfeeding women, due to potential risks to the fetus or infant.
* Inability or unwillingness to comply with the study protocol, including scheduled visits, tests, and procedures.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A cohort of 100 PBC patients treated with ursodiol and seladelpar
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
ALP and bilirubin levels | through study completion, up to 18 months
  Pruritus severity using the pruritus numeric rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Mangesh Pagadala, MD, Principal Investigator — Methodist Heath System

IPD SHARING:
Plan to Share IPD: No